CLINICAL TRIAL: NCT07045363
Title: Effectiveness of an Embedded Community-based Heart-Age Risk Education Model (E-CHARM) in Improving Cardiovascular Risk Awareness and Health Behaviors Among Older Adults With Hypertension: a Randomized Controlled Trial
Brief Title: Embedded Community-based Heart-Age Risk Education Trial in Cinese Primary Healthcare
Acronym: E-CHARM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke Kunshan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025HC064
Record Dates: First submitted 2025-06-09; First posted 2025-07-01 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Hypertension
Keywords: Heart Age; Health education
MeSH Terms: conditions — Hypertension; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Control Group) (No Intervention): Participants in this arm will receive standard hypertension management as per Chinese national guidelines, including regular follow-up with primary care physicians. They will not receive a Heart Age report or structured cardiovascular risk communication.
- Heart Age Communication (Intervention Group) (Experimental): Participants in this arm will receive a personalized Heart Age report based on their annual health check data (blood pressure, cholesterol, glucose, BMI, smoking). The report will be explained by the physician during the routine follow-up visit using a standardized script. The session lasts 3-5 minutes and is integrated into existing workflow.
  Interventions: Behavioral: Cognitive Intervention

INTERVENTIONS:
Behavioral: Cognitive Intervention — Participants in the intervention arm will receive a personalized one-page Heart Age report based on data from their government-funded annual health check. The report is delivered by trained physicians using a standardized communication script during a routine follow-up visit. The control group receives usual chronic disease care without structured risk communication.
  Arms: Heart Age Communication (Intervention Group)

SUMMARY:
This study evaluates the effectiveness of a brief Heart Age-based risk education intervention embedded in routine primary care for older adults with hypertension in China. The intervention uses routine health check data to generate a personalized one-page Heart Age report, delivered by physicians during regular follow-up visits. The trial tests whether this approach improves risk awareness and self-management behavior without disrupting clinical workflow.

DETAILED DESCRIPTION:
This is a randomized controlled trial conducted a community health center in Kunshan, Jiangsu, China. Approximately 600 older adults (≥60 years) with hypertension will be recruited following completion of their national annual health check. Participants will be randomized 1:1 to receive either standard care or a Heart Age report with a brief scripted explanation delivered during their next follow-up consultation. The primary outcome is change in cardiovascular risk awareness at 3 months. Secondary outcomes include behavior change(measured by questionnaires); implementation outcomes (feasibility, acceptability, fidelity) will be measured in the intervention group. Clinical indicators (e.g., blood pressure, glucose) will be extracted from health records at 12 months as exploratory outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥60 years
* Diagnosed with hypertension
* Completed their government-funded annual health check within the past 3 months
* Scheduled for a routine follow-up consultation within the enrollment window -Able to provide informed consent-

Exclusion Criteria:

* Diagnosed dementia or severe cognitive impairment
* Terminal illness
* Participation in another clinical intervention trial

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-07-19 (Estimated); Primary Completion 2025-10-20 (Estimated); Study Completion 2026-07-20 (Estimated)

PRIMARY OUTCOMES:
Change in cardiovascular disease (CVD) risk awareness | 3 months
  assessed using a 10-item CVD Knowledge Questionnaire adapted from the Chinese version of the Cardiovascular Disease Attitudes and Beliefs Questionnaire (ABCD-C) and the Heart Disease Fact Questionnaire (HDFQ). Each item is scored as 1 (correct) or 0 (incorrect/Don't know), yielding a total score range from 0 to 10. Higher scores indicate greater knowledge and awareness of CVD risk factors.

SECONDARY OUTCOMES:
Change in physical activity level | 3 months
  Change in self-reported physical activity level, measured using an 11-level categorical scale developed for this study and adapted from the WHO Stepwise approach. Responses range from 1 (completely inactive) to 11 (vigorous activity >25 miles/week or >8 hours/week). Higher scores indicate greater physical activity level.
Change in dietary behavior: fruit intake | 3 months
  Change in self-reported fruit consumption frequency, measured by the question: "On how many days per week do you usually eat fruit?" (0-7 days). Higher values indicate higher frequency of fruit intake.
Change in dietary behavior: table salt use | 3 months
  Change in self-reported table salt use, measured by a single item adapted from the WHO STEPS questionnaire: "Do you usually add salt or salty condiments (e.g., soy sauce) at the table?" Responses on a 5-point scale: 1 = Always, 5 = Never. Higher scores indicate lower frequency of adding table salt.
Change in medication adherence | 3 months
  Change in self-reported medication adherence, assessed using the Morisky Medication Adherence Scale, 4-item version (MMAS-4). Each item scored as Yes = 1, No = 0, for a total score range of 0-4. Lower scores indicate better medication adherence.
Implementation outcomes 1: Feasibility (intervention group only) | 3 months
  Measured using the Feasibility of Intervention Measure (FIM), 4 items, each scored on a 5-point Likert scale (1 = Strongly disagree, 5 = Strongly agree). Higher scores indicate greater perceived feasibility.
Implementation outcomes 2: Acceptability (intervention group only) | 3 months
  Measured using the Acceptability of Intervention Measure (AIM), 4 items, each scored on a 5-point Likert scale (1 = Strongly disagree, 5 = Strongly agree). Higher scores indicate greater acceptability.
Implementation outcomes 3: Fidelity (intervention group only) | 3 months
  Assessed using patient-reported and provider-reported delivery checks with categorical response options (e.g., explained fully, partially, not explained).

OTHER OUTCOMES:
Change in systolic blood pressure | 12 months
  Mean change in systolic blood pressure (mmHg) extracted from routine health records.
Change in diastolic blood pressure | 12 months
  Mean change in diastolic blood pressure (mmHg) extracted from routine health records.
Change in body mass index (BMI) | 12 months
  Mean change in body mass index (BMI, kg/m²) extracted from routine health records.
Change in fasting plasma glucose | 12 months
  Mean change in fasting plasma glucose level (mmol/L) extracted from routine health records.
Change in total cholesterol | 12 months
  Mean change in total cholesterol level (mmol/L) extracted from routine health records.
Change in low-density lipoprotein cholesterol (LDL-C) | 12 months
  Mean change in low-density lipoprotein cholesterol (LDL-C, mmol/L) extracted from routine health records.
Change in high-density lipoprotein cholesterol (HDL-C) | 12 months
  Mean change in high-density lipoprotein cholesterol (HDL-C, mmol/L) extracted from routine health records.
Change in triglycerides | 12 months
  Mean change in triglyceride level (mmol/L) extracted from routine health records.

CONTACTS AND LOCATIONS:
Overall Officials: Guanzhou Wang, Principal Investigator — Duke University
Locations (1):
- Tinglin Community Health Center, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
IPD will not be made publicly available due to data protection regulations and privacy concerns under local Chinese health authority guidelines. However, de-identified aggregated data may be shared upon reasonable request for academic research purposes. Requests should be submitted to the corresponding author and will be reviewed by the study steering committee.